CLINICAL TRIAL: NCT03460158
Title: Prospective Evaluation of Minimally Invasive Facial Cosmetic Procedures Through Measured Volumetric Changes and Patient Reported Outcomes
Brief Title: Prospective Evaluation of Facial Cosmetic Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 827003
Record Dates: First submitted 2017-09-15; First posted 2018-03-09 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cosmetic Techniques
Keywords: facial filler; Retylane; aesthetic improvement; volumizing fillers
MeSH Terms: interventions — Restylane-L

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Restylane-L®, Restylane-L® Lyft, and Restylane Silk® (Experimental): Hyaluronic acid
  Interventions: Drug: Restylane-L®; Drug: Restylane-L® Lyft; Drug: Restylane Silk®

INTERVENTIONS:
Drug: Restylane-L® — Restylane-L® for the indication for mid-to-deep dermal implantation for moderate to severe facial wrinkles and folds, such as nasolabial folds.
  Other Names: Hyaluronic acid gel
Drug: Restylane-L® Lyft — Restylane-L® Lyft is for the indication of implantation into the deep dermis to superficial subcutis for the correction of moderate to severe facial folds and wrinkles, such as nasolabial folds and malars (cheek/cheek bone area).
  Other Names: Hyaluronic acid gel
Drug: Restylane Silk® — Restylane Silk® is for the indication for submucosal implantation for lip augmentation and dermal implantation for correction of perioral rhytids in patients over the age of 21.
  Other Names: Hyaluronic acid gel

SUMMARY:
A prospective, trial to quantitatively and qualitatively compare the dermal fillers for the treatment of age related aesthetic changes.

DETAILED DESCRIPTION:
Dermal fillers have been approved for the treatment of age related aesthetic changes, including facial volume loss, and attenuation of the static and dynamic rhytid. Despite widespread use of volumizing fillers there is little data quantifying the subjective benefit of these minimally invasive treatments from the patient perspective. Furthermore, there is little data comparing the subjective benefit with true objective volumetric results. Such data will provide much needed information for patient counselling and treatment optimization for patient perceived outcomes.

This study is to determine the patient reported outcomes of three different dermal fillers and establish the volumetric changes over 90 days. Screening will be performed during the patient's office visit. Approximately 100 patients will be enrolled. Patients will participate up to 90 days (Day 1, 14 days, 28 days, and 90 days).

ELIGIBILITY:
Inclusion Criteria:

* Female patients 40 - 65 years of age

Exclusion Criteria:

* Male patients
* Prior surgical facial rejuvenation procedures
* Facelift
* Neck lift
* Blepharoplasty
* Facial fat grafting
* Prior minimally invasive rejuvenation procedure ≤ 12 months
* Known contraindications to devices or drugs used in this study
* Facial paralysis
* Congenital facial asymmetry
* Pregnant women
* Patient actively taking blood thinners

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivona Percec, MD,PhD, Principal Investigator — University of Pennsylvania Health System
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis HD, Mazzaferro D, Habarth-Morales TE, Messa CA 4th, Talwar AA, Desai AA, McAuliffe PB, Broach RB, Serletti JM, Percec I. A Large Prospective Volumetric and Patient-Reported Outcome Analysis of Hyaluronic Acid Facial Fillers. Plast Reconstr Surg. 2025 Oct 1;156(4):550-559. doi: 10.1097/PRS.0000000000012135. Epub 2025 Apr 1. PMID 40178806

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restylane-L®, Restylane-L® Lyft, and Restylane Silk®
Started | 101
Completed | 101
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Restylane-L®, Restylane-L® Lyft, and Restylane Silk®
Number analyzed (Participants) | 101
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53.2 [49.1 to 56.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American/Black | 8
  Race: Caucasian/White | 92
  Race: Asian | 1
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 24.4 [21.8 to 27.6]
Smoking History [Count of Participants; unit: Participants]
  Never | 62
  Current | 11
  Former | 27
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction With Validated FACE-Q Aesthetics Survey
Description: Absolute Change of the Patient Satisfaction using the validated FACE-Q Aesthetics questionnaire for patient reported assessment of treatment by domain.
  The absolute change from the patient reported outcome score prior to injection to the patient reported score immediate post-injection. Increase in numeric value indicates the larger patient reported improvement, except for psychosocial distress module where a decrease in numeric value indicates patient improvement. Maximum change 99 and Minimum Change 0.
Time Frame: 2 week post injections
Population: Subject who completed the validated patient reported FACE-Q Aesthetics survey 2 week post-injections
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Restylane-L®, Restylane-L® Lyft, and Restylane Silk®
Number analyzed (Participants) | 97
score on a scale
  Satisfaction with Facial Appearance. (Maximum change 99 and Minimum Change 0). | 28.0 [17.0 to 41.0]
  Aging Appraisal. (Maximum change 99 and Minimum Change 0). | 24.0 [8.5 to 41.5]
  Appraisal of Lines: Nasolabial Folds. (Maximum change 99 and Minimum Change 0). | 36.0 [12.0 to 58.0]
  Appraisal of Lines: Marionette Lines. (Maximum change 99 and Minimum Change 0). | 36.0 [19.0 to 58.0]
  Satisfaction with Lips. (Maximum change 99 and Minimum Change 0). | 23.5 [4.5 to 41.0]
  Satisfaction with Cheekbones. (Maximum change 99 and Minimum Change 0). | 32.0 [17.0 to 53.5]
  Satisfaction with Cheeks. (Maximum change 99 and Minimum Change 0). | 43.0 [23.0 to 60.0]
  Satisfaction with Lower Face and Jawline. (Maximum change 99 and Minimum Change 0). | 35.0 [20.0 to 55.0]
  Psychological Function. (Maximum change 99 and Minimum Change 0). | 13.0 [0.0 to 31.0]
  Social Function. (Maximum change 99 and Minimum Change 0). | 8.0 [0.0 to 29.0]
  Appearance-Related Psychosocial Distress. (Maximum change 99 and Minimum Change 0). | -12.0 [-29.0 to 0.0]

2. Secondary Outcome: Correlate Patient Satisfaction With Volumetric Measurements
Description: Linear correlation of relative volumetric change over relative patient satisfaction scale change. These values are reported as correlation coefficients and are unit less.
Time Frame: upto 90 days
Population: Patients who received Hyaluronic acid and patient reported outcomes (PRO)
Measure: Number (95% Confidence Interval); unit: correlation coefficient (unit less)
Arm/Group | Restylane-L®, Restylane-L® Lyft, and Restylane Silk®
Number analyzed (Participants) | 40
correlation coefficient (unit less)
  2 weeks post injection | 0.0226 [-0.2779 to 0.3232]
  4 weeks post injection | -0.1796 [-0.4691 to 0.1099]
  12 weeks post injection | -0.3692 [-0.5934 to -0.1451]
Statistical Analysis 1: Comparison: Restylane-L®, Restylane-L® Lyft, and Restylane Silk®; Two-sample t test with equal variances the null hypothesis is the relative change in volume and relative change in patient reported outcomes will be the same at 2 weeks post injection; Test type: Other; p = 0.8822, t-test, 2 sided; Mean Difference (Final Values) = 0.023, Standard Error of Mean 0.1524
Statistical Analysis 2: Comparison: Restylane-L®, Restylane-L® Lyft, and Restylane Silk®; Two-sample t test with equal variances the null hypothesis is the change in volume and change in patient reported outcomes will be the same at 4 weeks post injection; Test type: Other; p = 0.2223, t-test, 2 sided; Mean Difference (Final Values) = -0.180, Standard Error of Mean 0.1466
Statistical Analysis 3: Comparison: Restylane-L®, Restylane-L® Lyft, and Restylane Silk®; Two-sample t test with equal variances the null hypothesis is the change in volume and change in patient reported outcomes will be the same at 12 weeks post injection; Test type: Other; p = 0.0015, t-test, 2 sided; Mean Difference (Final Values) = -0.369, Standard Error of Mean 0.113

3. Secondary Outcome: Volumetric Changes of Treatment
Description: 3-dimensional photography to measure volumetric changes in each treatment
Time Frame: immediately post injection, 2 weeks, 4 weeks, and 12 weeks
Population: Volume Maintenance of Whole Face
Measure: Median (Inter-Quartile Range); unit: cc
Arm/Group | Restylane-L®, Restylane-L® Lyft, and Restylane Silk®
Number analyzed (Participants) | 99
cc
  post injection | 9.86 [7.37 to 12.6]
  2 weeks | 8.80 [6.30 to 11.0]
  4 weeks | 7.63 [5.85 to 10.6]
  12 weeks | 5.79 [3.20 to 9.38]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Restylane-L®, Restylane-L® Lyft, and Restylane Silk®
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT03460158/Prot_SAP_000.pdf